CLINICAL TRIAL: NCT05286060
Title: Open-label Phase II Trial for the Combination of GX-188E HPV DNA Vaccine With GX-I7 or Pembrolizumab OR the Triple Combination of GX-188E HPV DNA Vaccine, GX-I7, and Pembrolizumab in Patients With Advanced, Resectable HPV Type 16 or 18 Positive Head and Neck Cancer (Expanded Cohort)
Brief Title: Trial of the Combination of GX-188E Vaccination, GX-I7 and Pembrolizumab in Patients With Advanced, Resectable HPV Type 16 and/or 18 Positive Head and Neck Cancer
Acronym: GENUINE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yonsei University (Other)
Collaborators: Genexine, Inc. (Industry); NeoImmuneTech (Industry)
Responsible Party: Principal Investigator, Chang Gon Kim, Principal Investigator, Yonsei University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2021-1786
Record Dates: First submitted 2022-03-06; First posted 2022-03-18 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — efineptakin alfa; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- GX-188E 2mg, IM: 1st day of week 1, 2, and 4; GX-I7 1200㎍/kg (Experimental): IV:1st day of week 1 and 4, IV:1st day of week 1 and 4
  Triple combination of GX-188E HPV DNA Vaccine, GX-I7, and Pembrolizumab
  Interventions: Drug: GX-188E, GX-I7, Pembrolizumab
- GX-188E 2mg, IM: 1st day of week 1, 2, and 4; Pembrolizumab 200mg, IV:1st day of week 1 and 4 (Experimental): Combination of GX-188E HPV DNA Vaccine and Pembrolizumab as an Expanded Cohort
  Interventions: Drug: GX-188E, Pembrolizumab
- GX-188E 2mg, IM: 1st day of week 1, 2, and 4; GX-I7 360㎍/kg,GX-188E 2mg, (Experimental): IM: 1st day of week 1, 2, and 4; GX-I7 360㎍/kg, IM: 1st day of week 2; Pembrolizumab 200mg, IV:1st day of week 1 and 4
  Triple combination of GX-188E HPV DNA Vaccine, GX-I7, and Pembrolizumab as an Expanded Cohort
  Interventions: Drug: GX-188E, GX-I7, Pembrolizumab
- GX-188E 2mg, IM: 1st day of week 1, 2, and 4; GX-I7 360㎍/kg, IM: 1st day of week 2 (Experimental): Combination of GX-188E HPV DNA Vaccine and GX-I7 as an Expanded Cohort
  Interventions: Drug: GX-188E, GX-I7

INTERVENTIONS:
Drug: GX-188E, GX-I7, Pembrolizumab — Drug 1: GX-188E GX-188E, 2mg (1.0mg/0.5ml/vial), Intramuscular administration using electroporator Other Name: Tirvalimogene teraplasmid Drug 2: GX-I7 GX-I7 1200㎍/kg, intramuscular administration Other Name: NT-I7, rhIL-7-hyFc, efineptakin alfa Drug 3: Pembrolizumab pembrolizumab 200mg (100mg/4mL/vial), Intravenous administration Other Name: Keytruda®
  Arms: GX-188E 2mg, IM: 1st day of week 1, 2, and 4; GX-I7 1200㎍/kg
Drug: GX-188E, Pembrolizumab — Drug 1: GX-188E GX-188E, 2mg (1.0mg/0.5ml/vial), Intramuscular administration using electroporator Other Name: Tirvalimogene teraplasmid Drug 2: Pembrolizumab pembrolizumab 200mg (100mg/4mL/vial), Intravenous administration Other Name: Keytruda®
  Arms: GX-188E 2mg, IM: 1st day of week 1, 2, and 4; Pembrolizumab 200mg, IV:1st day of week 1 and 4
Drug: GX-188E, GX-I7, Pembrolizumab — Drug 1: GX-188E GX-188E, 2mg (1.0mg/0.5ml/vial), Intramuscular administration using electroporator Other Name: Tirvalimogene teraplasmid Drug 2: GX-I7 GX-I7 360㎍/kg, intramuscular administration Other Name: NT-I7, rhIL-7-hyFc, efineptakin alfa Drug 3: Pembrolizumab pembrolizumab 200mg (100mg/4mL/vial), Intravenous administration Other Name: Keytruda®
  Arms: GX-188E 2mg, IM: 1st day of week 1, 2, and 4; GX-I7 360㎍/kg,GX-188E 2mg,
Drug: GX-188E, GX-I7 — Drug 1: GX-188E GX-188E, 2mg (1.0mg/0.5ml/vial), Intramuscular administration using electroporator Other Name: Tirvalimogene teraplasmid Drug 2: GX-I7 GX-I7 360㎍/kg, intramuscular administration Other Name: NT-I7, rhIL-7-hyFc, efineptakin alfa
  Arms: GX-188E 2mg, IM: 1st day of week 1, 2, and 4; GX-I7 360㎍/kg, IM: 1st day of week 2

SUMMARY:
The study is open label, phase II clinical trial for the Combination of GX-188E HPV DNA Vaccine with GX-I7 or Pembrolizumab OR the Triple Combination of GX-188E HPV DNA Vaccine, GX-I7, and Pembrolizumab in Patients With Advanced, Resectable HPV Type 16 or 18 Positive Head and Neck Cancer.

DETAILED DESCRIPTION:
<Preoperative medication> [GX-188E 2mg: 1st day of week 1, 2, and 4; GX-I7 360㎍/kg or 1200㎍/kg: 1st day of week 2; Pembrolizumab 200mg: 1st day of week 1 and 4] Drug 1: GX-188E (Cohort I, II, III, IV) GX-188E, 2mg (1.0mg/0.5ml/vial), Intramuscular administration (IM) using electroporator Drug 2: GX-I7 (Cohort I, III, IV) GX-I7 360㎍/kg or 1200㎍/kg (Varies by cohort), intramuscular administration (IM) Drug 3: Pembrolizumab (Cohort I, II, III) pembrolizumab 200mg (100mg/4mL/vial), Intravenous administration (IV) <Operation> Surgery 2 to 8 weeks after completion of the test medication. <Posr OP CCRT> Physician's discretion

ELIGIBILITY:
[Inclusion Criteria]

1. A patient aged 19 or older at the time of signing the informed consent
2. Histologically identified, resectable local progressive, HPV positive (positive in p16 immunohistochemistry and positive in HPV-16 and/or HPV-18 nucleic acid tests) locally advanced (LA) head and neck squamous cell carcinoma (HNSCC) patients
3. A patient has never received other chemotherapy before the study
4. Eastern Cooperative Oncology Group (ECOG) performance status 0-1
5. Life expectancy of > 6 months
6. Patient agreed to provide storage tumor tissue samples or fresh biopsy samples for baseline biomarker tissue analysis including PD-L1 staining during biopsy or surgery must be present. If there is no storage tissue and there is no tumor lesion that can be sampled from biopsy or surgery, it will be excluded from the test.
7. Patients with suitable organ function. Samples must be collected within 28 days prior to the initiation of clinical trial drugs.
8. Patient with measurable diseases defined based on RECIST v.1.1.
9. For fertile woman (WOCBP), patient with negative results of serum or urine pregnancy tests conducted within 72 hours prior to the first administration of clinical trial drugs. If the urine test result is positive or cannot be confirmed negative, a serum pregnancy test should be performed.
10. Fertile woman must agree to use appropriate double contraception by 120 days after the entire course of this trial and the last administration of clinical trial drugs. Woman who are menopause (over 45 years of age and have no menstruation for more than a year) and women who are surgically infertile are exempt from this requirement.

    Note: abstinence is permitted if it is the daily lifestyle of the test subject and the contraceptive method preferred by the test subject.
11. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.

[Exclusion Criteria]

1. Unresectable metastatic or recurrent cancer.
2. Patients who are currently in progress or have been confirmed to have other malignant diseases that required active treatment within the past three years.

   Note: Subjects with skin basal cell carcinoma, skin squamous cell carcinoma, or in situ carcinoma (e.g., breast cancer) that have been treated for potential complete recovery purposes are not excluded.
3. Patients expected to require other forms of anti-neoplasm therapy during the test; This treatment includes systemic chemotherapy, radiation therapy, biotherapy, or immunotherapy not specified in the protocol.
4. Patients with a history of active central nervous system (CNS) metastasis and/or carcinoma meningitis.
5. Patients who have previously received treatment using anti-PD-1, anti-PD-L1, or anti-PD-L2 drugs or have received treatment using drugs directly acting on other irritating or co-inhibitory T cell receptors (e.g., CTLA-4, OX40, CD137).
6. Patients suffering from active autoimmune diseases requiring systemic immunosuppressive treatment (e.g., use of disease modulators, corticosteroids, or immunosuppressant) within the past two years. Alternative therapy (e.g., thyroxine, insulin, or physiological corticosteroid replacement due to adrenal or pituitary dysfunction) is not considered a form of systemic therapy and is therefore acceptable.
7. Patients who received homogeneous solid organ transplantation or homogeneous bone marrow transplantation.
8. Patients who have been administered non-PD-1/PD-L1/PD-L2, anti-cancer monoclonal antibodies (mAb, e.g., bevacizumab, cetuximab, etc.) within 4 weeks prior to the first administration of the clinical trial drug or have not yet recovered (e.g., grade 1 or baseline level).
9. Patients who received systemic chemotherapy including other clinical trial drugs within 4 weeks before the first administration of this clinical trial drug or received targeted hypogermic therapy with a half-life of less than 48 hours within 2 weeks.

   Note: The subject must have recovered to the baseline level or below in all adverse reactions caused by previous treatment. Neuropathy under grade 2 and/or anemia under grade 2 may be suitable.

   Note: If the subject has undergone major surgery, the subject must be properly recovered from toxicity and/or complications caused by the intervention prior to commencement of treatment.
10. Patients who had received radiation therapy within two weeks prior to the initiation of clinical trial drugs. The test subjects must have recovered from all radiation-related toxicity.
11. Patients who have transfused blood products (including platelets or red blood cells) within 4 weeks before the first administration of clinical trial drugs or have administered colony stimulation factors (Includes G-CSF, GM-CSF, or recombinant red blood cell generators).
12. Patients with bilateral hydronephrosis that cannot be alleviated by ureteral stent or percutaneous renal fistula formation.
13. Patients with severe (≥3) hypersensitivity to one of the additive components of study drugs.
14. Patients with a history of (non-infectious) interstitial pneumonia requiring steroids or currently suffers from interstitial pneumonia.
15. Patients diagnosed with immunodeficiency or patients receiving long-term systemic steroid therapy (dose exceeding 10 mg of prednisone per day) or receiving other immunosuppressive treatments in any form within 7 days prior to the first administration of clinical trials.
16. Patients with risk factors for intestinal obstruction or intestinal perforation (e.g., acute diverticulitis, intraabdominal abscess, and abdominal carcinoma, but not limited).
17. Patients who are currently participating in clinical trials for other clinical trial drugs or have participated in the past have received clinical trial treatment or used clinical trial devices within 4 weeks before the first administration of this clinical trial drug.

    Note: If more than 4 weeks have elapsed since the last administration of the previous clinical trial drug, subjects who have entered the follow-up stage of the clinical trial may participate in this trial.
18. Unstable/Inadequate heart function:

    * Symptomatic ischemia
    * Unregulated or clinically significant abnormal conduction (e.g., ventricular tachycardia during antiarrhythmia treatment); 1-degree ventricular block or asymptomatic LAFB/RBBB is suitable
    * Cardiomyopathy within the past 6 months
    * Congestion Heart failure (New York Heart Association III - IV grade
19. Active infected patients who need systemic treatment.
20. Patients with confirmed human immunodeficiency virus (HIV) infection, and/or hepatitis B or C history, or hepatitis B surface antigen (HBsAg)/ hepatitis B virus (HBV) DNA or hepatitis C antibody or RNA test positive. Active hepatitis C is defined as a case where Hep CAb results are positive and quantitative HCV RNA results are found to be higher than the lower detection limit of the analysis.
21. Patients with a history of active tuberculosis.
22. Patients who received a live vaccine within 30 days before the first administration of the clinical trial drug. Examples of live vaccines include, but are not limited to, the following: Measles, mumps, rubella, pox/shingles, yellow fever, rabies, BCG, and typhoid vaccines. Seasonal flu vaccines used in injections are generally viral vaccines, but nasal flu vaccines (e.g., Flumist®) are not allowed because they are weakly poisoned vaccines.
23. Patients who have been confirmed to have mental illness or substance abuse that may interfere with their ability to cooperate with the requirements of this test.
24. A patient who transplanted an implantation electronic device (e.g., a pacemaker) into the body.
25. Fertile women with positive urine pregnancy test results (e.g., within 72 hours) prior to administration of clinical trial drugs. If the urine test is positive or has not been confirmed negative, a serum pregnancy test is required.
26. Pregnant or lactating patients.
27. Patients who are likely to confuse the test results or interfere with the subject's participation in the entire duration of the test. Patients who have a history of abnormalities in conditions, treatments, laboratory tests, or currently have such evidence, regardless of type, where participation in clinical trials is judged to be in the best interest of the subjects.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Major pathologic response | Immediately after the surgery
  Evaluate the pathologic response in resected tumor tissue. The major pathologic response is defined as less than 10% viable tumors after treatment.

SECONDARY OUTCOMES:
Radiologic response | Immediately after the surgery
  Based on Response Evaluation Criteria in Solid Tumors 1.1
Safety | UP to 5years
  Based on the National Cancer Institute Common Terminology Criteria, version 5.0
Pathologic complete response | Right after the surgery. Up to 5 years
  Defined as no residual viable tumor in the surgically resected specimen.
Locoregional recurrence-free survival | UP to 5years
  Time from surgical resection to locoregional recurrence
Distant recurrence-free survival | UP to 5years
  Time from surgical resection to distant recurrence
Recurrence-free survival | UP to 5years
  Time from surgical resection to any type of recurrence
Disease-free survival | UP to 5years
  Time from surgical resection to locoregional recurrence, distant recurrence, or death from any cause, whichever occurred first
Overall survival | Up to 5years
  Time from date of treatment initiation to the date of death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Hye Ryun Kim, Principal Investigator — Severance Hospital
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No